CLINICAL TRIAL: NCT02181114
Title: Computer Tailored Education Program to Reduce Disparities in Living Donor Kidney Transplant
Brief Title: Your Path to Transplant: A Randomized Control Trial of A Tailored Computer Education Intervention for Living Donor Kidney Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Amy D. Waterman, Director, Patient Engagement, Diversity, and Education, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DK088711-1; NCT01553864 (obsolete NCT alias)
Record Dates: First submitted 2014-06-27; First posted 2014-07-03 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: End Stage Renal Disease
Keywords: Coaching; Educational Materials; Expert System; Living Donor Kidney Transplant
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Expert System Coaching (Experimental): Patients in the intervention group will receive coaching based off the answers provided in the computer-based Expert System that is designed to track their readiness level to pursue a living donor kidney transplant.
  Interventions: Behavioral: Expert System Coaching
- Control (No Intervention): Patients in the control group will only receive the standard of care education that is offered at the UCLA Kidney and Pancreas Transplant Center which consists of a powerpoint presentation on their Evaluation Day appointment.

INTERVENTIONS:
Behavioral: Expert System Coaching — Patients will receive coaching and feedback over the phone and stag-appropriate educational materials (i.e. paphlets, brochures, personalized feedback report) based on their answers to the survey questions and where they are in their kidney transplant evaluation process.
  Arms: Expert System Coaching

SUMMARY:
Because of the deceased donor organ shortage, more kidney patients are considering whether to receive kidneys from family and friends, a process called living donor kidney transplantation (LDKT). Although Blacks are 3.4 times more likely to develop end stage renal disease, they are less likely to receive LDKTs. To address this disparity, this randomized controlled trial will assess whether Black and White transplant patients' knowledge and receipt of LDKTs can be increased when they receive access to the Your Path to Transplant computerized Expert System (YPT). This trial will also examine how other known patient, family, and healthcare system barriers to LDKT impact YPT's effectiveness.

Nine hundred (900) Black,White and Hispanic ESRD patients presenting for transplant medical evaluation at University of California-Los Angeles Kidney and Pancreas Transplant Program (UCLA-KPTP) in Los Angeles, California will be stratified by race and randomly assigned to one of two education conditions (YPT vs. Usual Care Education). As they undergo transplant evaluation, patients in the YPT condition will receive individually-tailored feedback reports, coaching, and socioeconomic resource guidance associated with reducing barriers to access to LDKT. Control patients will receive usual care transplant education provided by UCLA-KPTP. Changes in knowledge, readiness to pursue LDKT, pros/cons to LDKT, and self-efficacy will be assessed at four time points: prior to presenting at the transplant center (baseline), during transplant evaluation (approximately 2 months post-baseline), and 4- and 8-months post-baseline. Completion of transplant evaluation and receipt of LDKTs will be assessed 18-months post-baseline.

At the conclusion of the study, we will have developed an innovative and cost-effective YPT Computerized Expert System that could be utilized to tailor LDKT discussion and education in different medical settings based on the needs of individual patients of different races.

DETAILED DESCRIPTION:
This longitudinal, parallel randomized control trial has two treatment conditions with equal allocation, the YPT intervention and the standard of care transplant education as provided by UCLAKPT. Patients in both groups will be assessed at four time points: 1) a phone survey at baseline; 2) a phone survey at 4 months post-baseline; 3) a phone survey at 8 months post-baseline; and 4) a medical records review at 4, 8 and 18 months post-baseline. Additionally, patients in the YPT intervention group will receive individualized YPT transplant education at various time points: 14 days post-baseline by phone, the in-person transplant education (ITE) session, during the 4 month post-baseline survey, and during the 8 month post-baseline survey. The date of the ITE education session cannot be fixed because it may occur at different points in each patient's transplant evaluation process.

As patient records are received via the transplant database, a data manager will determine which are eligible for the study, then assign eligible patients a PIN that has been pre-randomized to treatment group before uploading the record to the recruitment database. Randomization will be completed by using a computer software program called TTMX (Transtheoretical Model Expert). Knowledge of treatment assignment is required at and after this stage so that the YPT expert system can be delivered to patients randomized to the intervention condition. Patients will be randomized into one of two groups: usual care or intervention group.

Usual Care Control Group-UCLA The control group for this trial consists of the usual care for transplant education which, for this facility, begins when a referral is made. A physician, patient medical group or dialysis center can make the referral. Once UCLAKPTP receives the patient's information via a patient information form and their insurance has been verified, the patient is called to schedule an Education Seminar and a one-on-one evaluation appointment. Next, both UCLAKPTP mail out an "Appointment Letter" for the patient to complete and bring with them to Evaluation Day. These packets include a UCLAKPTP Appointment Letter and a Doctor's Information Worksheet. Patients are asked to fill out and bring the Information Worksheet with them on their appointment day. The evaluation day is a full day of group education, physician appointment, meetings with several coordinators of care and if necessary completing several medical tests with blood and urine collection. During the two hour group education a power point presentation is given that reviews different transplantation options including living and deceased donors as well as high risk donors. The social worker concludes the education by reviewing important insurance information with the group. Next, the patients have a series of individual appointments with the transplant physician (either a nephrologist or a surgeon), a social worker and the transplant coordinator where they can ask questions and will receive additional information on transplant. Psychosocial evaluations are completed by the social workers to identify any risk factors or red flags which would contradict transplant as a treatment. This routine is standard for all patients evaluated for transplant. Patients in this group will be surveyed at baseline, 4 months and 8 months post baseline. These surveys will be conducted over the phone and can last up to 50 minutes each.

YPT Intervention Group Patients in the intervention group with receive individualized YPT transplant education at four time points. Their total participation is estimated to be 2.5 hours. Printed materials and videos will be sent to the patients after each time point. Patients will also receive individualized feedback reports based on their stage of readiness to pursue DDKT and LDKT. In addition to being tailored to the individual's stage of readiness, these reports will address any concerns the patient has mentioned as well as answers to knowledge questions the patient may have missed.

YPT intervention: baseline time point. We will first administer verbal consent form and assess for ineligibility criteria. After consent has been given and eligibility determined, we will conduct a baseline assessment of the patient's demographics, knowledge, decision making, readiness, and self-efficacy for both DDKT and LDKT. Family support and living donor availability will also be assessed for LDKT. This time point is estimated to last 40 minutes. At the end of the survey the patient will be asked schedule a time to conduct the first education session.The education session will occur at any time up to 14 days after the baseline assessment and will last between 20-30 minutes. The coach will then discuss the patient's readiness to pursue DDKT. This will be guided by the patient's stage of change. Next, the coach addresses the benefits of DDKT and provides coaching for any concerns the patient mentioned in the assessment. After this, the coach will discuss the patient's over all confidence for pursuing DDKT and then provide itemized feedback for problems the patient believes will prevent them from pursuing DDKT. The coach will then provide the same education and coaching for LDKT. At the end of the education session the coach will inform the patient that they will meet the patient on the day of their ITE.

The coach will then mail a folder containing the first set of educational materials which includes factsheets, brochures and the patient's personalized, tailored feedback report.

YPT intervention: ITE time point. The ITE session will occur at the UCLAKPTP during the patient's medical evaluation visits. It is expected to last 40 minutes. Patients will be taken to a semi-private area in the transplant center at either facility and re-assess the patient's readiness to pursue DDKT and LDKT as well as the perceived benefits and concerns. The patient's confidence for pursuing both DDKT and LDKT will also be re-assessed. We will provide feedback to the patient based on any changes in readiness, confidence, and perceived benefits or concerns that may have occurred since the initial assessment. DDKT feedback will occur directly after DDKT re-assessment and LDKT feedback will occur after LDKT re-assessment. The patient will then be asked to watch a 10 minute video while we print off the patient's personalized feedback report. Based on the patient's stage of change, one of two videos will be shown: "Pursuing Donation" to those patients who are in the pre-contemplation and contemplation phases and "Exploring Donation" will be for patients in all of the other stages. At the end of the session we will give the patient a second folder with educational materials, a DVD, and their personalized feedback report.

YPT intervention: 4 month and 8 month time point. We will contact the patient four months and eight months after their baseline survey. Pre-survey reminder postcards will be sent one month prior to the survey. It is estimated that each survey will last 45 minutes. These interviews will be similar to the baseline survey given at the beginning of the trial. However, we will not re-assess demographic information, comorbidities, or unmet needs. At both time points, we will provide tailored feedback throughout the interview. This will occur immediately after the re-assessment of potential barriers to pursuing transplant, knowledge, and transplant decision making for both DDKT and LDKT. During the eight month interview, we will ask the patient questions regarding the cultural competency of their medical providers, their decision about which treatment to pursue, and their ability to have made an informed decision as to whether or not pursue DDKT or LDKT. As with previous time points, individualized feedback reports and tailored education will be sent to the patients following the phone call.

YPT patients: 4, 8, and 18 month medical record review. Patients' medical records will be reviewed at 4, 8 and 18 months after their baseline survey in order to determine whether they had: 1) been waitlisted for transplant; 2) received a DDKT; 3) received an LDKT; 4) gone inactive or been determined ineligible for transplant; 5) died.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black, White, or Hispanic
* Must not have been deemed kidney transplant ineligible by UCLA Kidney and Pancreas Transplant Program
* Cannot be listed at another transplant center
* Can read English

Exclusion Criteria:

* Does not self-identify as Black, White, or Hispanic
* Deemed ineligible to receive a kidney transplant by UCLA Kidney and Transplant Program
* Listed at another transplant center
* Cannot read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 815 (Actual)
Dates: Start 2014-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Patient LDKT Attitude & Decision-Making Measure: Readiness | up to 8 months post-Baseline
  Using validated measures, patients will be asked how ready they are to get a DDKT by reporting whether they are "not considering getting a DDKT in the next six months" (Precontemplation), "considering getting a DDKT in the next six months" (Contemplation), "preparing to get a DDKT in the next 30 days" (Preparation), "undergoing evaluation to get a DDKT" (Action) or "listed and waiting to get a DDKT" (Maintenance). Patients will also be asked how ready they are to pursue LDKT and to rate whether they are "not considering taking actions in the next six months to pursue LDKT" (Precontemplation), "considering taking actions in the next six months to pursue LDKT" (Contemplation), "preparing to take actions in the next 30 days to pursue LDKT" (Preparation), or "taking actions to pursue LDKT" (Action).

SECONDARY OUTCOMES:
Patient LDKT Attitude & Decision Making Measure: Decisional Balance | up to 8 months post-Baseline
  Decisional Balance measures will assess how patients weigh the relative importance of possible LDKT and DDKT positive and negative outcomes (e.g., "My living donor will feel good seeing my health improve"). Patients will be asked to rate the importance of each statement on a 5-point scale ranging from, (1) "Not important" to (5) "Extremely important".
Patient LDKT Attitude & Decision Making Measure: Self-efficacy | up to 8 months post-Baseline
  The Self-Efficacy scale measures the confidence an individual has in his/her ability to pursue transplant in a wide variety of challenging situations (e.g., "If your friends and family were unsupportive of you getting a transplant") on a scale from (1) "Not at all confident" to (5) "Completely confident".
Patient LDKT Attitude & Decision Making Measure: Small Steps towards LDKT and DDKT | up to 8 months post-Baseline
  To assess their steps toward transplant, patients will be asked to respond whether they have "Already done", "Are planning to do", or "Don't plan to do" a list of actions related to LDKT and DDKT. Examples of steps toward LDKT include "Read information/watch videos about getting a living donor transplant" and "Ask potential donors to be tested", while examples of steps toward DDKT include "Share educational materials about deceased donation with people in your life" and "Follow-up with the transplant coordinator until transplant evaluation is complete".
Patient LDKT Attitude & Decision Making Measure: Transplant Knowledge | up to 8 months post-Baseline
  Patients will be asked 11 true/false and 8 multiple choice questions to determine their level of knowledge regarding basic facts, advantages, risks and outcomes of DDKT and LDKT (e.g., "Patients older than 80 years can receive transplants"; "Compared to transplants from donors who have died, how long do transplants from living donors last?"). A measure of transplant knowledge is then created by summing the number of correct answers to the questions.
Final Outcome: Pursuit of Transplant | 18 months post-Baseline
  Finally, patients' electronic medical records at UCLA and data from the Scientific Registry for Transplant Recipients (SRTR) will be reviewed 18 months post-baseline to create a final study outcome for each patient. At the study's conclusion, the patient will be coded as to: 1) be waitlisted for a DDKT; 2) have received a DDKT; 3) have received a LDKT; 4) have been determined to be medically ineligible for transplant; 5) have died; or 6) have dropped out of evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Waterman, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA Division of Nephrology, Los Angeles, California
  - University of Rhode Island, Kingston, Rhode Island

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Waterman AD, Peipert JD, Cui Y, Beaumont JL, Paiva A, Lipsey AF, Anderson CS, Robbins ML. Your Path to Transplant: A randomized controlled trial of a tailored expert system intervention to increase knowledge, attitudes, and pursuit of kidney transplant. Am J Transplant. 2021 Mar;21(3):1186-1196. doi: 10.1111/ajt.16262. Epub 2020 Sep 15. PMID 33245618
- [Derived] Waterman AD, Robbins ML, Paiva AL, Peipert JD, Kynard-Amerson CS, Goalby CJ, Davis LA, Thein JL, Schenk EA, Baldwin KA, Skelton SL, Amoyal NR, Brick LA. Your Path to Transplant: a randomized controlled trial of a tailored computer education intervention to increase living donor kidney transplant. BMC Nephrol. 2014 Oct 14;15:166. doi: 10.1186/1471-2369-15-166. PMID 25315644